CLINICAL TRIAL: NCT05653544
Title: Natural History and Longitudinal Clinical Assessments in a Spanish Cohort of Primary Mitochondrial Myopathies
Brief Title: Natural History in Primary Mitochondrial Myopathies
Acronym: NHPMM
Status: Recruiting | Type: Observational
Sponsor: Cristina Domínguez González (Other)
Responsible Party: Sponsor-Investigator, Cristina Domínguez González, Cristina Domínguez González, MD, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Other Study IDs: 22/493
Record Dates: First submitted 2022-11-29; First posted 2022-12-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Primary Mitochondrial Myopathies
Keywords: mtDNA; TK2; large scale single deletion; multiple deletions; POLG; TWNK

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — DNA, muscle biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mitochondrial myopathy: Mitochondrial myopathy, confirmed genetically

SUMMARY:
This is a longitudinal study in a cohort of patients with a genetic diagnosis of Primary Mitochondrial Myopathy to describe the natural history of the disease and identify clinical, biochemical, molecular, and radiological variables that allow evaluation of the severity and progression of the disease and may be useful in future clinical trials.

DETAILED DESCRIPTION:
Mitochondrial Diseases (MD) are among the most frequent inherited metabolic diseases. Despite their high impact on patients, there are still no authorized drugs capable of modifying their clinical course. MD are clinically and genetically heterogeneous disorders, with muscular symptoms being one of their main manifestations. When muscular symptoms predominate, the disorder is classified as a Primary Mitochondrial Myopathy. In recent years, there have been significant advances in developing potential new treatments in this field. However, the absence of natural history studies makes the design and interpretation of clinical trials difficult and leads to long delays or even failures in the development of new treatments. The investigators propose to characterize in-depth a cohort of patients with Primary Mitochondrial Disorders due to mutations in the mitochondrial DNA (mtDNA) or in genes located in the nuclear genome (nDNA), from a clinical perspective but also a radiological, biochemical, and molecular point of view, and carry out a longitudinal follow-up of these parameters to identify those that are better correlated with severity and that allow measuring changes in the patient's clinical situation. With this objective, the investigators will analyze clinical variables (evaluation of motor function through manual force exploration, functional scales, and timed test, quality of life scales, serum biomarkers (growth differentiation factor 15 (GDF15) and fibroblast growth factor 21 (FGF21)), levels of heteroplasmy for cases harboring mtDNA mutations and mtDNA copy-number, and muscle magnetic resonance image of the lower extremities with quantification of fat replacement. All parameters will be evaluated at the beginning of the study and then annually during two years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Muscle symptoms: exercise intolerance and fatigue, myalgia, recurrent rhabdomyolysis, chronic progressive external ophthalmoplegia and/or muscular weakness
* Primary mtDNA mutation or pathogenic mutations in nDNA, especially in genes related to mtDNA maintenance such as TK2, POLG, TWNK and RRM2B, among others.

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Primary Mitochondrial Myopathy with a genetic diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor Function (endurance) | 36 months
  6 minute walking test (6MWT)

SECONDARY OUTCOMES:
Motor Function (functional scale) | 36 months
  North Star Ambulatory Assessment (NSAA)
Biomarkers | 36 months
  Analysis of levels of GDF15 y FGF21 annually
Levels of heteroplasmy | 36 months
  Analysis of levels of heteroplasmy annually
Muscle magenitc resonance image (MRI) | 36 months
  Quantification of the fat fraction in muscle MRI, annually

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario 12 Octubre, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dominguez-Gonzalez C, Hernandez-Voth A, de Fuenmayor-Fernandez de la Hoz CP, Guerrero LB, Moris G, Garcia-Garcia J, Muelas N, Leon Hernandez JC, Rabasa M, Lora D, Blazquez A, Arenas J, Martin MA. Metrics of progression and prognosis in untreated adults with thymidine kinase 2 deficiency: An observational study. Neuromuscul Disord. 2022 Sep;32(9):728-735. doi: 10.1016/j.nmd.2022.07.399. Epub 2022 Jul 16. PMID 35907766
- [Background] Dominguez-Gonzalez C, Fernandez-Torron R, Moore U, de Fuenmayor-Fernandez de la Hoz CP, Velez-Gomez B, Cabezas JA, Alonso-Perez J, Gonzalez-Mera L, Olive M, Garcia-Garcia J, Moris G, Leon Hernandez JC, Muelas N, Servian-Morilla E, Martin MA, Diaz-Manera J, Paradas C. Muscle MRI characteristic pattern for late-onset TK2 deficiency diagnosis. J Neurol. 2022 Jul;269(7):3550-3562. doi: 10.1007/s00415-021-10957-0. Epub 2022 Mar 14. PMID 35286480
- [Background] Bermejo-Guerrero L, de Fuenmayor-Fernandez de la Hoz CP, Serrano-Lorenzo P, Blazquez-Encinar A, Gutierrez-Gutierrez G, Martinez-Vicente L, Galan-Davila L, Garcia-Garcia J, Arenas J, Muelas N, Hernandez-Lain A, Dominguez-Gonzalez C, Martin MA. Clinical, Histological, and Genetic Features of 25 Patients with Autosomal Dominant Progressive External Ophthalmoplegia (ad-PEO)/PEO-Plus Due to TWNK Mutations. J Clin Med. 2021 Dec 22;11(1):22. doi: 10.3390/jcm11010022. PMID 35011763
- [Background] Rodriguez-Lopez C, Garcia-Cardaba LM, Blazquez A, Serrano-Lorenzo P, Gutierrez-Gutierrez G, San Millan-Tejado B, Muelas N, Hernandez-Lain A, Vilchez JJ, Gutierrez-Rivas E, Arenas J, Martin MA, Dominguez-Gonzalez C. Clinical, pathological and genetic spectrum in 89 cases of mitochondrial progressive external ophthalmoplegia. J Med Genet. 2020 Sep;57(9):643-646. doi: 10.1136/jmedgenet-2019-106649. Epub 2020 Mar 11. PMID 32161153